CLINICAL TRIAL: NCT06117566
Title: A Phase Ib/IIa Study to Evaluate the Safety and Preliminary Efficacy of WX390 Combined With Toripalimab in Patients With Advanced Solid Tumors
Brief Title: A Study of WX390 Combined With Toripalimab in Patients With Advanced Solid Tumors
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Jiatan Pharmatech Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JYP0390M203
Record Dates: First submitted 2023-10-30; First posted 2023-11-07 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Solid Tumor
MeSH Terms: interventions — toripalimab

STUDY DESIGN:
Intervention Model Description: WX390 continuous oral dosing (0.5 mg once a day) WX390 continuous oral dosing (0.7 mg once a day) WX390 continuous oral dosing (0.9 mg once a day) Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks)
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- WX390 0.5 mg + Toripalimab 240mg (Experimental): Participants will receive WX390 continuous oral dosing (0.5 mg once a day) and Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks).
  Interventions: Drug: WX390; Drug: Toripalimab
- WX390 0.7 mg + Toripalimab 240mg (Experimental): Participants will receive WX390 continuous oral dosing (0.7 mg once a day) and Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks).
  Interventions: Drug: WX390; Drug: Toripalimab
- WX390 0.9 mg + Toripalimab 240mg (Experimental): Participants will receive WX390 continuous oral dosing (0.9 mg once a day) and Toripalimab fixed dose (240mg, intravenous, Day 1, every 3 weeks).
  Interventions: Drug: WX390; Drug: Toripalimab

INTERVENTIONS:
Drug: WX390 — WX390 tablet, once a day
  Other Names: WXFL10030390
Drug: Toripalimab — 240 mg, Day 1, every 3 weeks

SUMMARY:
The goal of this clinical trial is to evaluate the safety and preliminary efficacy of WX390 combined with Toripalimab in patients with advanced solid tumors. The main questions it aims to answer are:

* the maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) of WX390;
* safety and preliminary in combined therapy. Participants will be treated with WX390 orally and Toripalimab intravenously, and follow the efficacy and safety evaluation according to the protocol.

DETAILED DESCRIPTION:
This study will be an open-label, multicenter phase Ib/IIa clinical trial. After being informed about the study and potential risks, all patients giving written informed consent will undergo a 4-week screening period to determine eligibility for study entry. And then patents will be administered for 8 cycles treatment and 8 weeks safety follow up after the last dose of treatment. The efficacy and safety measures will be conducted and collected every cycle.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years of age
* Histological or cytological confirmed advanced solid tumor, standard regimen failed or no standard regimen available
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Life expectancy of more than 3 months
* At least one measurable lesion according to RECIST 1.1
* Adequate organ function，
* Signed and dated informed consent

Exclusion Criteria:

* Anti-cancer therapy within 30 days prior to the initiation of investigational treatment
* Major surgery within 30 days prior to the initiation of study treatment
* Received corticosteroids treatment or other immunodepressant within 2 weeks before the first dose of study treatment
* Toxicity from a previous anti-tumor treatment that does not return to Grade 0 or 1 (except for alopecia)
* Patients who are suffering active interstitial lung disease
* Evidence of ongoing or active serious infection
* History of human immunodeficiency virus (HIV) infection or active hepatitis B or C infection
* Inability to take medication orally
* Abuse of alcohol or drugs
* People with cognitive and psychological abnormality or with low compliance
* Pregnant or lactating women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-11-18 (Actual); Primary Completion 2025-11-09 (Estimated); Study Completion 2025-11-09 (Estimated)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) and dose-limiting toxicity (DLT) in DLT observation period | up to 24 weeks
  The safety and tolerability of WX390 will be evaluated based on adverse events data. Other safety parameters include physical examination, clinical laboratory tests including coagulation function, renal function, hepatic function, blood glucose and blood lipid, etc.
Progression-free survival rate (PFS rate) | up to 24 weeks
  PFS rate: is defined as the proportion of patients without objective tumor progression or death.
Objective response rate (ORR) | up to 24 weeks
  ORR: is defined as the proportion of patients with complete response (CR) and partial response (PR) according to RECIST 1.1.

SECONDARY OUTCOMES:
Progression-free survival (PFS) | up to 48 weeks
  PFS: is defined as the time from randomization until objective tumor progression or death, whichever occurs first.
Overall survival (OS) | up to 48 weeks
  OS: is defined as the time from randomization until death from any cause.
Disease-control rate (DCR) | up to 24 weeks
  DCR: is defined as the proportion of patients with complete response (CR), partial response (PR) and stable disease (SD) according to RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Ding, PhD, Principal Investigator — the first affiliated hospital of Jilin university
Locations (1):
- the first affiliated hospital of Jilin university, Changchun, Jilin, China